CLINICAL TRIAL: NCT01788098
Title: Rheumatoid Arthritis Susceptibility Genes in Austrian and Slovak Population
Brief Title: Genetics and Mechanisms of Rheumatoid Arthritis
Acronym: RASGENAS
Status: Completed | Type: Observational
Sponsor: Slovak Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Stefan Zorad, Head of Laboratory, Slovak Academy of Sciences
Other Study IDs: RASGENAS; ATMOS N00024 (Other Grant/Funding Number: Cross Border Cooperation Slovakia - Austria 2007 - 2013)
Record Dates: First submitted 2013-02-03; First posted 2013-02-11 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Rheumatoid Arthritis; Leukocytes, Mononuclear; Genetic Association Studies
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — frozen immune cells frozen serum frozen DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rheumatoid Arthritis: Patients with rheumatoid arthritis
- Healthy controls: Healthy control subjects

SUMMARY:
The study is aimed at revealing genetic background in rheumatoid arthritis (RA). For that purpose samples of DNA will be collected from 500 RA patients and similar number of controls from whole Slovakia. Variations in several genes associated with RA will be evaluated. The second aim is to assess functional changes in immune cells from selected patients and their evaluation together with genetic background. The project has observational character without any intention to change the treatment of RA patients.

ELIGIBILITY:
Inclusion Criteria:

* rheumatoid arthritis or healthy

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis and healthy controls from Slovakia and Austria
Sampling Method: Probability Sample
Enrollment: 790 (Actual)
Dates: Start 2009-10; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Genetic association | 1 day
  Association of selected single nucleotide polymorphisms with rheumatoid arthritis.

SECONDARY OUTCOMES:
Peripheral blood mononuclear cells reactivity | 1 day
  Reactivity and functional changes of peripheral blood mononuclear cells obtained from patients with rheumatoid arthritis in comparison to healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Imrich, Study Chair — Slovak Academy of Sciences, Center for Molecular Medicine
Locations (1):
- Slovak Academy of Sciences, Center for Molecular Medicine, Bratislava, Slovakia